CLINICAL TRIAL: NCT03986879
Title: Relationship of the Intensity of Physical Activity Practice and Its Different Domains With Cardiac Autonomic Modulation in Adult Individuals
Brief Title: Relationship of the Physical Activity Practice and Its Different Domains With Cardiac Autonomic Modulation
Status: Completed | Type: Observational
Sponsor: Bruna Thamyres Ciccotti Saraiva (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Bruna Thamyres Ciccotti Saraiva, Clinical Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Organization: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Other Study IDs: 72191717.9.0000.5402
Record Dates: First submitted 2019-05-30; First posted 2019-06-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Adult Disease
Keywords: Physical Activity; Cardiovascular Health; Epidemiological
MeSH Terms: conditions — Disease; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Overall objective: To analyze the relationship of the physical activity practice measured directly with the autonomic cardiac modulation in adults. Specific objectives: i) to verify through the Baecke questionnaire whether the different domains of physical activity (work, leisure and occupational activities) are related in the same way to the autonomic cardiac modulation; ii) Analyze whether high blood pressure and resting heart rate values are related to poor cardiac autonomic modulation regardless of nutritional status.

DETAILED DESCRIPTION:
Cardiovascular disease is a major public health problem and has contributed to a high mortality rate in the adult population. One of the precursors of these diseases is low cardiac autonomic modulation. Thus, factors that may be related to greater cardiac autonomic modulation should be investigated with the aim of preventing cardiovascular diseases. One of these factors that may contribute to increases in cardiac autonomic modulation is the practice of physical activity. However, the studies investigating this relationship have been controversial, generally evaluating the practice of physical activity in a subjective way, and there is no clarity as to whether the different domains of physical activity would be related differently to cardiac autonomic modulation. Overall objective: To analyze the relationship of the physical activity practice measured directly with the autonomic cardiac modulation in adults. Specific objectives: i) to verify through the Baecke questionnaire whether the different domains of physical activity (work, leisure and occupational activities) are related in the same way to the autonomic cardiac modulation; ii) Analyze whether high blood pressure and resting heart rate values are related to poor cardiac autonomic modulation regardless of nutritional status. Implications: The results of this study will contribute to clarify the relationship between physical activity practice and cardiac autonomic modulation considering a large sample of subjects (n = 252), as well as whether the different domains of physical activity are related to autonomic modulation cardiac. These results may help in the elaboration of health promotion strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* be resident of the city of Anastácio-SP (Brazil)
* sign the informed consent form

Exclusion Criteria:

* use less than 5 valid accelerometer days
* present an error in heart rate variability greater than 5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will be composed of adults aged 18 years or older from the city of Santo Anastácio-SP located in the southeastern region of Brazil.
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic modulation | through study completion, an average of 1 year
  The heart rate variability will be collected by means of the POLAR V800.
Physical activity level - objective measure | through study completion, an average of 1 year
  Will be collected 7 days of accelerometry by ActiGraph's triaxial accelerometer wGT3X-BT giving the measure in counts per minute.

SECONDARY OUTCOMES:
Self-reported physical activity level questionnaire | through study completion, an average of 1 year
  Physical activity in different domains will be evaluated by the Baecke et al. (1982). This instrument evaluates the practice of physical activity through 16 questions in the last twelve months, considering the physical effort at work, the practice of sports activities or systematized exercises in leisure and leisure activities. At the end, this instrument offers a dimensionless score for each of the domains and the sum of the score of the three domains also determines the total amount of physical activity practiced by each of the evaluated individuals.
Systolic Blood pressure | through study completion, an average of 1 year
  The systolic blood pressure will be measured by means of the omron digital oscillometric device.
Diastolic Blood pressure | through study completion, an average of 1 year
  The diastolic blood pressure will be measured by means of the omron digital oscillometric device.
Self-reported practice of physical activity in childhood and adolescence | through study completion, an average of 1 year
  To evaluate the practice of physical activity in childhood (age 7 to 10 years) and adolescence (11-17 years) two questions will be asked: if they practiced some kind of sport in these phases of life with supervision of a teacher, with two alternatives of answer: yes or no.
Resting Heart Rate | through study completion, an average of 1 year
  The resting heart rate will be measured by means of the omron digital oscillometric device.
Body Mass | through study completion, an average of 1 year
  Individuals will be evaluated barefoot wearing light clothing. Body mass will be measured by means of a digital scale (Plenna, Brazil)
Height | through study completion, an average of 1 year
  Individuals will be evaluated barefoot wearing light clothing. The height will be evaluated by a fixed stadiometer on the wall.
Body Mass Index | through study completion, an average of 1 year
  The body mass index (BMI) will be calculated by dividing the body mass by the square of the height. Individuals classified up to 24.99 kg/m² will be considered as normal weight, those classified as having a BMI varying from 25.00 kg/m² up to 29.99 kg/m² will be classified as overweight and those with BMI ≥ 30 kg/m² as obese.
Waist Circumference | through study completion, an average of 1 year
  The waist circumference will be evaluated by an inextensible tape (Sanny, Brazil) and will consider the smallest circumference between the last rib and the iliac crest. Abdominal obesity will be considered in men with waist circumference ≥102 cm and women at 88 cm, following the recommendations of the World Health Organization (WHO, 1997).

CONTACTS AND LOCATIONS:
Overall Officials: Diego GD Christofaro, PhD, Principal Investigator — Universidade Estadual Paulista - UNESP
Locations (1):
- Diego Giulliano Destro Christofaro, Presidente Prudente, São Paulo, Brazil

REFERENCES:
- [Derived] Tebar WR, Ritti-Dias RM, Mota J, Saraiva BTC, Damato TM, Delfino LD, Farah BQ, Vanderlei LCM, Christofaro DGD. Relationship of Cardiac Autonomic Modulation with Cardiovascular Parameters in Adults, According to Body Mass Index and Physical Activity. J Cardiovasc Transl Res. 2021 Oct;14(5):975-983. doi: 10.1007/s12265-021-10101-3. Epub 2021 Jan 22. PMID 33483920
- [Derived] Tebar WR, Ritti-Dias RM, Saraiva BTC, Gil FCS, Delfino LD, Damato TMM, Aguilar BAS, Silva SCB, Mota J, Vanderlei LCM, Christofaro DGD. The relationship between physical activity intensity and domains with cardiac autonomic modulation in adults: An observational protocol study. Medicine (Baltimore). 2019 Oct;98(41):e17400. doi: 10.1097/MD.0000000000017400. PMID 31593091